CLINICAL TRIAL: NCT02332811
Title: An Open Label, Dose Titration Study of Sevelamer Carbonate Tablets & Powder in Hyperphosphatemic Chronic Kidney Disease Patients
Brief Title: An Open Label, Dose Titration Study of Sevelamer Carbonate Tablets & Powder in Hyperphosphatemic CKD Patients
Acronym: TOSCANA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVCARB10012; U1111-1160-6394 (Other: UTN)
Record Dates: First submitted 2014-12-16; First posted 2015-01-07 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Renal Failure Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CKD patients not on dialysis 800 mg (Experimental): Sevelamer carbonate 800 mg in tabs 3 times per day with meals
  Interventions: Drug: sevelamer carbonate 800mg
- CKD patients not on dialysis 2.4 g (Experimental): Sevelamer carbonate 2.4 g powder carbonate per day
  Interventions: Drug: sevelamer carbonate 2.4 g
- CKD patients on dialysis 800 mg (Experimental): Sevelamer carbonate 800 mg in tabs 3 times per day with meals
  Interventions: Drug: sevelamer carbonate 800mg
- CKD patients on dialysis 2.4 g (Experimental): Sevelamer carbonate 2.4 g powder carbonate per day
  Interventions: Drug: sevelamer carbonate 2.4 g

INTERVENTIONS:
Drug: sevelamer carbonate 800mg — Pharmaceutical form:tablet
  Route of administration: oral
  Other Names: Renvela
  Arms: CKD patients not on dialysis 800 mg; CKD patients on dialysis 800 mg
Drug: sevelamer carbonate 2.4 g — Pharmaceutical form:powder
  Route of administration: oral
  Other Names: Renvela
  Arms: CKD patients not on dialysis 2.4 g; CKD patients on dialysis 2.4 g

SUMMARY:
Primary Objective:

Evaluate the reduction in serum phosphorus from baseline to end of study with Sevelamer carbonate tablets 800 mg and Sevelamer carbonate Powder 2.4 g in chronic kidney disease (CKD) patients both on haemodialysis and not on dialysis

Secondary Objective:

Evaluate the safety on the basis of adverse events, changes in laboratory values and vital signs from baseline (Day 0) to Day 56 (End of treatment/ End of Study)

DETAILED DESCRIPTION:
10 weeks including, 2 weeks wash-out period and 8 weeks study treatment period

ELIGIBILITY:
Inclusion criteria :

Men or women 18 years of age or older suffering from CKD not on dialysis or on a stable haemodialysis regimen

* If currently on phosphate binder(s), willing to stop this and enter a 2 week washout period
* Willing to avoid any intentional changes in diet such as fasting or dieting
* Have the following laboratory measurement:

  * iPTH ≤ 1000 pg/mL at screening (including results obtained within 60 days prior to screening)
  * If not taking a phosphate binder, a serum phosphorus measurement >5.5 mg/dL (1.78 mmol/L) at Screening (Visit 1).
  * If taking a phosphate binder at screening, a serum phosphorus measurement > 5.5 mg/dL (1.78 mmol/L) after the two-weeks washout period at Visit 1a (Day 0).
* Willing and able to take Sevelamer carbonate alone as a phosphate binder for the duration of the study
* Willing and able to avoid antacids and phosphate binders containing aluminum, magnesium, calcium or lanthanum for the duration of the study
* Willing and able to maintain screening doses of vitamin D, and/or cinacalcet for the duration of the study, except for safety reasons
* If female and childbearing potential (pre-menopausal and not surgically sterile), willing to use an effective contraceptive method throughout study, which includes barrier methods, hormones, or intrauterine devices
* For patients not on dialysis expecting not to initiate dialysis for the duration of this study
* Signed informed consent
* Has not participated in any other investigational drug studies within 30 days prior to enrollment
* Level of understanding and willingness to cooperate with all visits and procedures as described by the study personnel

Exclusion criteria:

* Active dysphagia or swallowing disorder
* Predisposition or current bowel obstruction,
* Severe gastrointestinal (GI) motility disorders including severe constipation
* Active ethanol or drug abuse, excluding tobacco use
* Use of anti-arrhythmic or anti-seizure medications for arrhythmia or seizure disorders.
* In the opinion of the investigator, patient has poorly controlled diabetes mellitus, poorly controlled hypertension, active vasculitis, HIV infection, or any clinically significant unstable medical condition
* Planned renal transplant or parathyroidectomy within 3 months of Visit 1
* Pregnant or breast-feeding
* Evidence of active malignancy except for basal cell carcinoma of the skin
* Unable to comply with the requirements of the study
* Known hypersensitivity to sevelamer or any constituents of the study drug
* Any other condition, which in the opinion of the investigator will prohibit the patient's inclusion in the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The reduction in serum phosphorus from baseline to end of study with Sevelamer carbonate tablets 800 mg and Sevelamer carbonate Powder 2.4 g in chronic kidney disease (CKD) patients both on haemodialysis and not on dialysis | up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Russia, Moscow, Russia